CLINICAL TRIAL: NCT05905887
Title: A Phase 2 Study of Paclitaxel Plus Rivoceranib in Patients With GIST With a High P-glycoprotein Expression After Failure With at Least Imatinib, Sunitinib and Regorafenib
Brief Title: Rivoceranib Plus Paclitaxel in Patients With Gastrointestinal Stromal Tumor
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Hee Ryu, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC2301
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — apatinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rivoceranib plus paclitaxel (Experimental)
  Interventions: Drug: Rivoceranib Mesylate, Paclitaxel

INTERVENTIONS:
Drug: Rivoceranib Mesylate, Paclitaxel — Paclitaxel will be administered at 80mg/m2/day every four weeks at Day 1, Day 8 and Day 15 per cycle. One cycle consists of 4 weeks (28 days).
  Rivoceranib 400 mg orally once a day.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rivoceranib and paclitaxel combination therapy in patients with P-glycoprotein overexpressing GIST who failed standard treatment with imatinib, sunitinib, and regorafenib.

DETAILED DESCRIPTION:
With the development of KIT mutation and KIT tyrosine kinase inhibitor imatinib (GlivecTM, Novartis), survival of patients with advanced and/or metastatic gastrointestinal stromal tumor (GIST) has significantly improved. Recently, sunitinib (SuteneTM, Pfizer) and regorafenib (StivargaTM, Bayer) have been proven to be effective as second- and third-line treatment, respectively in GIST patients who failed to imatinib treatment. However, almost all patients eventually experience disease progression due to the development of drug resistance to first-line imatinib, second-line sunitinib treatment, and third-line regorafenib. As a fourth-line treatment, ripretinib was proven to prolong progression-free survival as compared to placebo with a median progression-free survival of 6.3 months in the Phase 3 INVICTUS study. However, ripretinib is not available in many regions including Korea, making it difficult to use. Therefore, a new treatment options are needed in the clinical setting post-imatinib, sunitinib and regorafenib.

Historic data suggest that GISTs do not respond to conventional cytotoxic chemotherapy, but systematic unbiased screening has not been performed. A recent large-scaled chemotherapy susceptibility screening with GIST cells showed that among a total of 89 chemotherapies, 37 have anti-cancer effect in at least one type of GIST cells. It was suggested that of these agents, transcriptional inhibitors and chemotherapies such as topoisomerase II, paclitaxel, and bortezomib would be effective. Based on these results, our group has recently performed a phase II study for evaluating efficacy and safety of paclitaxel in patients with advanced and/or metastatic GIST after failure of at least imatinib and sunitinib. Although paclitaxel showed overall limited anti-tumor efficacy, it was more effective in patients with low P-glycoprotein expression. Based on these study results, it was hypothesized that paclitaxel would also be effective in GIST patients, and a phase II study was conducted to evaluate the efficacy and safety of paclitaxel in 25 patients with advanced and/or metastatic GIST who failed imatinib and sunitinib treatment. At week 16, the disease control rate (DCR; response + stable lesion) was 16.7%, showing a limited anticancer effect. However, in patients with a low level of P-glycoprotein expression, the DCR was 25% at 16 weeks, suggesting that paclitaxel may be efficacious in this clinical setting. Subsequently, a phase II clinical trial of paclitaxel is currentl ongoing in patients with metastatic or progressive GIST with low P-glycoprotein expression who have failed imatinib, sunitinib, and regorafenib treatment in patients with a low P-glycoprotein expression level. However, data from Asan Medical Center suggest that only about 20% of GISTs have a low P-glycoprotein expression level (IHC score 3 points or less) in this clinical setting.

P-glycoprotein is a plasma membrane protein that acts as an efflux pump for drugs and is implicated in multidrug resistance. In particular, hydrophobic chemotherapeutic agents such as paclitaxel are known to be substrates of P-glycoprotein, supporting the concept that GIST patients with high P-glycoprotein expression may be resistant to paclitaxel. This raise the possibility that paclitaxel-based combination treatment may be considered when the function of P-glycoprotein is inhibited.

Ricoveranib is a mutikinase inhibitor with anti-angiogenic activity. In a phase 3 study conducted in China, rivoceranib improved overall survival compared to placebo as a 3rd-line treatment for metastatic gastric cancer. In addition, an improvement in progression-free survival compared to placebo was confirmed in the multinational phase 3 ANGEL study. Recently, the combination therapy of rivoceranib and camrelizumab, an immune checkpoint inhibitor, in unresectable liver cancer has been proven to improve survival results compared to sorafenib. When it comes to the treatment of GIST, the anti-angiogenic activity and inhibition of P-glycoprotein by rivoceranib suggest its potential use in GIST patients. In particular, when used in combination with paclitaxel in GIST whose P-glycoprotien expression level is high, rivoceranib is expected to have an additional or synergistic anti-tumor activity. In a phase 1 clinical study of metastatic gastric cancer, the combination therapy of rivoceranib and palclitaxel was confirmed to be safe as well as showing clinical efficacy. The recommended dose for phase 2 study was rivoceranib 400mg and paclitaxel 80mg/m2 (days 1,8 and 15, 4-week cycle).

The objective of this study is to evaluate the safety and efficacy of paclitaxel in combination with rivoceranib in patients with metastatic or advanced GIST with a high P-glycoprotein expression level after failure of at least imatinib, sunitinib and regorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older, at the time of acquisition of informed consent
* Histologically confirmed metastatic and/or advanced GIST with CD117(+), DOG-1(+), or mutation in KIT or PDGFRα gene
* P-glycoprotin IHC score > 3 (Tumor tissue with disease progression after regorafenib treatment)
* Failed (progressed and/or intolerable) after prior treatments for GIST, including at least imatinib and sunitinib, regorafenib.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 ~ 2
* Resolution of all toxic effects of prior treatments to grade 0 or 1 by NCI-CTCAE version 5.0
* At least one measurable lesion as defined by RECIST version 1.1.
* Adequate bone marrow, hepatic, renal, and other organ functions Neutrophil >1,500/mm3 Platelet > 100,000/mm3 Hemoglobin >8.0 g/dL Total bilirubin < 1.5 x upper limit of normal (ULN) AST/ALT < 2.5 x ULN Creatinine <1.5 x ULN
* Life expectancy > 12 weeks
* Washout period of previous TKIs or chemotherapy for more than 4 times the half life ((Imitinib and regorafenib need 1 week and sunitinib need 2 weeks.)
* Provision of a signed written informed consent

Exclusion Criteria:

* Women of child-bearing potential who are pregnant or breast feeding
* Women or men who are not willing to use effective contraception entering the study period or until at least 3 months after the last study drug administration.
* If any of the following applies within ≤ 6 months prior to starting study enrollment : Myocardial Infarction, severe instable angina, coronary/peripheral bypass, NYHA class III or IV congestive heart failure, stroke or transient ischemic attack, treatment required severe arrhythmia.
* Uncontrolled infection
* Acute and chronic liver disease and all chronic liver impairment.(But Patients with stable chronic hepatitis B are eligible)
* Uncontrolled gastrointestinal toxicities with toxicity greater than NCI CTCAE grade 2
* Acute, or chronic medical or psychiatric condition or laboratory abnormality such as active uncontrolled infection that difficult to study participation in the judgment of the investigator
* The patient experienced any bleeding episode considered life-threatening, or any grade 3 or 4 bleedig event. (required transfusion or endoscopic or surgical intervention)
* Currently clinically significant (within 7 days prior to screening) treatment of anticoagulants or other thrombolytic agents. A maximum dose of 325 mg/day of aspirin is allowed
* History of uncontrolled hypertension (blood pressure ≥140/90 mmHg and change in antihypertensive medication within 7 days prior to screening) that is not well managed by medication and the risk of which may be precipitated by a VEGF inhibitor therapy.
* History of clinically serious opearation, bone fracture or non-healing wounds within the last 3 weeks prior to screening
* History of other significant cardiovascular diseases or vascular diseases, within the last 6 months prior to screening (e.g., hypertensive crisis, and hypertensive encephalopathy or transient ischemic attack or significant peripheral vascular diseases] that, in the investigator's opinion, may pose a risk to the patient on VEGFR inhibitor therapy.
* History of clinically significant glomerulonephritis, biopsy-proven tubulointerstitial nephritis, crystal nephropathy, or other renal insufficiencies
* Known diagnosis of HIV infection (HIV testing is not mandatory).
* History of another primary malignancy that is currently clinically significant or currently requires active intervention.
* Patients with clinically suspected brain metastasis symptom, brain metastases as assessed by radiologic imaging
* Alcohol or substance abuse disorder.
* Known hypersensitivity to rivoceranib or any component of its formulation or history of severe hypersensitivity to including Cremophor R EL(polyoxyethylated castor oil) drug
* Concomitant treatment with strong inhibitors or inducers of CYP3A4, CYP2C9 and CYP2C19
* Active bacterial infections

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No